CLINICAL TRIAL: NCT01087424
Title: Phase II Study of Mini-CHOP Plus Rituximab in Non Previously Treated Patients Aged Over 80 Years With CD 20+ Diffuse Large B-Cell Lymphoma
Brief Title: Mini-CHOP and Rituximab in Patients Aged Over 80 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNH03-7B
Record Dates: First submitted 2009-08-26; First posted 2010-03-16 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R mini CHOP (Experimental): Induction : 3 cycles every 3 weeks Consolidation :3 cycles every 3 weeks
  Interventions: Drug: R mini CHOP

INTERVENTIONS:
Drug: R mini CHOP — Prednisone 40 mg/m2 D1 D2 D3 D4 D5 Rituximab 375 mg/m2 D1 Doxorubicine 25 mg/m2 D1 Cyclophosphamide 400 mg/m2 D1 Vincristine 1 mg/m2 D1

SUMMARY:
The purpose of the study is to evaluate efficacy and safety of R-miniCHOP for elderly patients with diffuse large B-Cell lymphoma (DLBC) Lymphoma aged over 80 years by measuring the overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven CD20+ diffuse large B-cell lymphoma (WHO classification). DLBCL with some small cell infiltration in bone marrow or lymph node may be included.
* Aged over 80 years.
* Ann Arbor stage I bulky, II, III or IV
* Age-adjusted International Prognostic Index equal to 0, 1, 2 and 3.
* Patient non previously treated.
* ECOG performance status ≤ 2.
* With a minimum life expectancy of 3 months.
* Negative HIV, HBV and HCV serologies test ≤ 4 weeks (except after vaccination).
* Having previously signed a written informed consent

Exclusion Criteria:

* Any other histological type of lymphoma.
* Any history of treated or non-treated indolent lymphoma.
* Central nervous system or meningeal involvement by lymphoma.
* Contra-indication to any drug contained in the chemotherapy regimens.
* Any serious active disease (according to the investigator's decision).
* Poor renal function (creatinin level>150µmol/l), poor hepatic function (total bilirubin level>30mmol/l, transaminases>2.5 maximum normal level) unless these abnormalities are related to the lymphoma.
* Poor bone marrow reserve as defined by neutrophils <1.5 G/l or platelets <100 G/l, unless related to bone marrow infiltration.
* Any history of cancer during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.
* Adult patient under tutelage.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Evaluating efficacy of R-miniCHOP by overall survival | 2 years overall survival

SECONDARY OUTCOMES:
Evaluating R-miniCHOP efficacy by Event free survival | 2 years event free survival

REFERENCES:
- [Derived] Ghesquieres H, Larrabee BR, Haioun C, Link BK, Verney A, Slager SL, Ketterer N, Ansell SM, Delarue R, Maurer MJ, Fitoussi O, Habermann TM, Peyrade F, Dogan A, Molina TJ, Novak AJ, Tilly H, Cerhan JR, Salles G. FCGR3A/2A polymorphisms and diffuse large B-cell lymphoma outcome treated with immunochemotherapy: a meta-analysis on 1134 patients from two prospective cohorts. Hematol Oncol. 2017 Dec;35(4):447-455. doi: 10.1002/hon.2305. Epub 2016 Jun 10. PMID 27282998
- [Derived] Copie-Bergman C, Cuilliere-Dartigues P, Baia M, Briere J, Delarue R, Canioni D, Salles G, Parrens M, Belhadj K, Fabiani B, Recher C, Petrella T, Ketterer N, Peyrade F, Haioun C, Nagel I, Siebert R, Jardin F, Leroy K, Jais JP, Tilly H, Molina TJ, Gaulard P. MYC-IG rearrangements are negative predictors of survival in DLBCL patients treated with immunochemotherapy: a GELA/LYSA study. Blood. 2015 Nov 26;126(22):2466-74. doi: 10.1182/blood-2015-05-647602. Epub 2015 Sep 15. PMID 26373676
- [Derived] Peyrade F, Jardin F, Thieblemont C, Thyss A, Emile JF, Castaigne S, Coiffier B, Haioun C, Bologna S, Fitoussi O, Lepeu G, Fruchart C, Bordessoule D, Blanc M, Delarue R, Janvier M, Salles B, Andre M, Fournier M, Gaulard P, Tilly H; Groupe d'Etude des Lymphomes de l'Adulte (GELA) investigators. Attenuated immunochemotherapy regimen (R-miniCHOP) in elderly patients older than 80 years with diffuse large B-cell lymphoma: a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2011 May;12(5):460-8. doi: 10.1016/S1470-2045(11)70069-9. Epub 2011 Apr 7. PMID 21482186